CLINICAL TRIAL: NCT04591847
Title: Pregnancy Outcomes and Vitamin D Level Among Vitamin D Supplementation During Pregnancy : A Double-blind Randomized Placebo Controlled Trial
Brief Title: Pregnancy Outcome and Vitamin D Level Among Vitamin D Supplementation During Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 121/2563
Record Dates: First submitted 2020-09-14; First posted 2020-10-19 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy Outcome Among Vitamin D Supplementation During Pregnancy
Keywords: Vitamin D; 25-hydroxyvitamin D; Pregnancy; Infant
MeSH Terms: interventions — Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D supplemented group (Experimental): Vitamin D2 20000 IU 1 tab oral weekly start at GA 18 -22 weeks until delivery
  Interventions: Drug: Vitamin D 2
- Placebo group (Experimental): Placebo drug (Appearance same as Vitamin D2) 1 tab oral weekly start at GA 18 -22 weeks until delivery
  Interventions: Drug: Placebo drug

INTERVENTIONS:
Drug: Vitamin D 2 — Vitamin D2 20000IU 1 tab oral weekly
  Arms: Vitamin D supplemented group
Drug: Placebo drug — Placebo drugs 1 tab oral weekly
  Arms: Placebo group

SUMMARY:
To compared pregnancy outcome (Serum vitamin D level in mother and infant , preeclampsia rate, preterm birth rate, Infant birth weight, Infant length , APGAR score) between pregnant women who were given vitamin D supplementation and pregnant women who were given placebo

ELIGIBILITY:
Inclusion Criteria:

* Thai female
* Singleton pregnancy
* Age at 18 years old or more
* Gestational age at 18-22 weeks
* Accept to enroll

Exclusion Criteria:

* Pregnant women who not planned to delivery at Rajavithi hospital
* Abnormal kidney function
* Use antiepileptic drugs , or vitamin D supplementation
* Allergy to vitamin D
* Who were diagnosed as vitamin D deficiency

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Serum 25-OH vitamin D level in pregnant women | At delivery time
  measure in nmol/L
Serum 25-OH vitamin D level in umbilicalcord blood | At delivery time
  measure in nmol/L

SECONDARY OUTCOMES:
Preeclampsia | During pregnancy until delivery
  Measure by clinical and laboratory of preeclampsia
  ้high blood pressure ( >= 140/90 mmHg) with proteinuria (UPCI > 0.3 mg/dL or Urine protein 24 hours > 300 mg) or in absence of proteinuria with new onset of any of the following
  * thrombocytopenia : Platelet count less than 100,000 x 10^9 /L
  * Serum creatinine > 1.1 mg/dL or doubling of the serum creatinine
  * Elevated liver transaminases to twice normal
  * Pulmonary edema
  * New onset headache unresponsive to medication
  * Visual symptom
Preterm birth | At delivery time
  Delivery before GA 37 weeks
Infant APGAR score | At delivery time
  Measure at delivery time score 10/10
  Appearance : Cyanotic, pale all over = 0 , Peripheral cyanotic only = 1 , Pink = 2 Pulse : 0 bpm = 0 , <100 = 1, 100-140 = 2 Grimace : no response to stimulation = 0 , Grimace(facial movement ,weak cry) = 1 Cry when stimulated = 2 Activity (tone) : floppy = 0 , Some flexion = 1 , Well flexed and resisting extension = 2 Respiration : Apnoeic = 0 , Slow irregular = 1 , Strong cry = 2
Infant birth weight | At delivery time
  measure in kilograms
Infant length | At delivery time
  measure in centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi hospital, Bangkok, Thailand